



### NON SUBSTANTIAL AMENDMENT

N° 1 Amendment No. **FINAL** Version No.

PM1541 Study Code 2015-002877-40

EudraCT n°

8th March 2017 Date

# A MULTICENTRE, RANDOMIZED, DOUBLE-BLIND, PARALLEL-GROUP, CONTROLLED STUDY, TO ASSESS THE EFFICACY AND SAFETY OF P-3074 CUTANEOUS SPRAY, SOLUTION, IN THE TREATMENT OF MALE PATTERN BALDNESS

## **Sponsor:**

Polichem SA,

50 Val Fleuri Luxembourg,

hereby legally represented by its branch located in:

Lugano-Pazzallo CH-6912 (Switzerland), Via Senago, 42 D

Tel. +41-91-986.40.00

Fax +41-91-986.40.01

## Centres affected by the amendment:

All the centres involved in the study

## CONFIDENTIALITY STATEMENT:

This confidential document is the property of Polichem S.A. The recipient agrees that no unpublished information contained herein may be disclosed without the prior written approval of Polichem S.A.

## AMENDMENT APPROVAL FORM

PROTOCOL No.: PM541

**PROTOCOL TITLE:** A MULTICENTRE, RANDOMIZED, DOUBLE-BLIND, PARALLEL-GROUP, CONTROLLED STUDY, TO ASSESS THE EFFICACY AND SAFETY OF P-3074 CUTANEOUS SPRAY, SOLUTION, IN THE TREATMENT OF MALE PATTERN BALDNESS

DATE OF ISSUE: Non Substantial Amendment 1 - Final Version - 8th March 2017

| | PPD | |
|------------------------|------------|------|
| PPD | PPD | PPD |
| Polichem S.A. | Signature | Dáte |
| | PPD | PPD |
| PPD | PPD | PPD |
| Polichem S.A. | Signature | Date |
| COUNTRY: | | |
| Principal Investigator | | |
| Printed Name | Signature | |
| I I IIIICU I Vallic | Digitature | Date |

These signatures constitute approval of this protocol amendment and provide the necessary assurance that this study will be conducted according to all stipulations of the amendment.

## RATIONALE FOR NON-SUBSTANTIAL AMENDMENT

This non-substantial amendment concerns the increasing of the screening period, initially planned in the study protocol, as 1 week  $\pm$  3 days. After the signature of the Informed Consent Form by patient, the severity of the baldness condition has to be evaluated by a global photography of the scalp, made by the Study Blind Assessor. However, before sending the photos to the Blind Assessor, a quality check has to be performed by the Image Company responsible of this study, aimed at detecting potential exposure errors, the presence of oil/wet on the hair or hair combing style leading the photo not evaluable. In case of the occurrence of any of these issues, the Image Company may ask for a reshooting of the target baldness area, prolonging in this way the screening period and leading to an out of window visit. Therefore, due to this technical period of evaluation, the Sponsor decided to have 2 weeks  $\pm$  5 days as screening period. For this reason, and following the European Directive 2010/C 82/01 with regards to a minor increase in the duration of the trial (< 10 % of the overall time of the trial), the Sponsor decided to implement this protocol change as not-substantial.

Other minor clarifications, comments, text deletions, typo corrections and a general adjustment to the protocol, not impacting on the safety or physical or mental integrity of the clinical trial participants, or the scientific value of the trial, have been included in this not-substantial amendment.

Therefore, the Sponsor submits the below consolidated protocol versions reflecting the aforementioned changes:

- Protocol PM1541 Version 4.0, track changes and clean dated 8<sup>th</sup> March 2017

In the same context, the Sponsor notifies the update of the Investigator's Brochure, Version 6 dated 17 Feb 2017 and the EudraCT form with the change of the legal representative and the change of the company's name of Therametrics Clinical Supply Services Srl into Euromed Clinical Supply Services Srl (enclosed also the authorization of the Italian Authority).

The most relevant sections changed are displayed below, with corrections/additions/deletions in red bold text. The same changes will be applied throughout the document.

| Ta | h | A | Λf | co | ní | en | te |
|-----|-------|---|-----|----|----|----|----|
| - 4 | . , , | | .,, | | | | |

The pages' numbers were updated.

| Synopsis |
|---|
| Experimental Design: |
| omissis |
| the site for reshoot until the images are considered evaluable. |
| omissis |
| Study Procedures |
| Seven clinical examinations are planned for each patients, as follows: |
| - Screening, Visit 1 (Week -1 2) |
| Statistical Methods |
| omissis |
| The variance-covariance matrix of unstructured form will be used in order to model the correlation, within |
| each patient, between the three two repeated measurements (over the post-baseline visits). |
| omissis. |
| The secondary efficacy variables, MHGQ scores, Blind assessor and local investigator assessments of |
| patient hair growth/loss, will be analysed using the same mixed linear model for repeated measures (MMRM) employed for the analysis of primary efficacy data. |
| (MINIKINI) employed for the analysis of primary efficacy data. |
| Study Protocol |
| 2.2 Secondary end-points |
| omissis |
| For the purpose of assessment of changes in hair growth by investigators and blind assessor, |
| screening visits (where global photos are taken) will act as baseline. |
| 3.2 Randomization |
| omissis |
| In the same context, patients have to take in 1 mg tablet oral finasteride (or its placebo) daily until the |
| end of a 24-week treatment course (Visit 6). |
| omissis |
| 2.2 Diindina |
| 3.3 Blinding |

The randomization list will be generated by IXRS vendor and implemented in IXRS system. Additionally, IXRS vendor will generate treatment kit number list that will be provided to the drug supply vendor for the preparation of the treatment kits.

Two (2) copies of the list are generated and securely provided as follows:

- **→** one copy is sent to the manufacturer for the preparation of the individual treatment boxes
- > one copy is sent to the IXRS vendor for management of drug supply and emergency unblinding.

| Neither the members of the clinical unit nor the CPL or the CRA/monitor will have access to the |
|---|
| randomisation eode data or to the treatment kit number list. Upon DB lock, the randomization file |
| will be transferred to CRO for analysis all subjects will be unblinded through IXRS. |
| omissis |

# 3.3.1 Emergency code and unblinding procedures ....omissis... The Investigator will be able to break the blind for an individual patient via IXRS according to the unblinding procedure or via code envelope supplied with each treatment kit. ...omissis.

# 3.5 Study flow-chart

| | Screening | | Tre | eatment Pha | se | | Follow up Phase (End of Study) | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|
| Visit | Visit 1 | Random<br>Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | |
| | -Weeks 12 | Day 1±35d | Week<br>4±3d | Week<br>8±3d | Week<br>12±3d | Week<br>24±3d | Week 28±3d | |
| Patient's Informed<br>Consent Form signature | X | | | | | | | |
| Demographic and habits information | X | | | | | | | |
| Physical examination§ | X | | | | | X | X | X |
| Medical history/current diseases | X | | | | | | | |
| Prior and concomitant medication | X | | | | | | | |
| Vital signs | X | | | | | X | X | X |
| Check all<br>Inclusion/exclusion<br>criteria | X | X | | | | | | |
| Enrolment | X | | | | | | | |
| Dispense patient's card | X | | | | | | | |
| Global Photograph | X | <u>X*</u> | | | X | X | | X |
| Investigator assessment | X* | | | | X | X | | X |
| Blind Assessor (entry eligibility) | X | | | | | | | |
| Blind Assessor (efficacy) | X* | | | | X | X | | X |
| Safety Laboratory examinations | X | | | X | | X | | X |
| Check record concomitant medication | | X | X | X | X | X | X | X |

| CCI | | | | | | | |
|---|---|---|---|---|---|---|---|
| Macrophotography (hair count) | X | | | X | X | | X |
| MHGQ Questionnaire | | | | X | X | | X |
| Sexual Dysfunction<br>Questionnaire (IIEF-2) | | X | X | X | X | X | X |
| Randomization | X | | | | | | |
| Dispense study medication | X | | | X | | | |
| Collect / return study medication | | X# | X <sup>#</sup> | X | X | | X |
| <b>Drug Application at site</b> | | X | X | X | X | | |
| Drug Compliance | | | | X | X | | X |
| Dispense study diary to the patient | X | | | | | | |
| Check of patient's study diary | | X | X | X | X | X | X |
| Collect / return study diary | | | | | | X | X |
| Severity score for skin irritation | | X | X | X | X | X | X |
| Record AEs | X | X | X | X | X | X | X |

<sup>\*</sup> Reshoot of global photograph if required \* Assessment of hair growth will be performed by investigator and blinded assessor at visits 5 and 6/EOT using global photographs as baseline

<sup>#</sup> Due to the blood samplings for PK/PD analyses, the patients have to bring with them the study drug also at Visits 3 and 4, for an administration on site

<sup>§</sup> Height will be measured only at screening

## 5.1 Study visits and procedures

....omissis.....

MaximumThe study duration will be 29 about 30 weeks. A written informed consent will be obtained before any study assessment or procedure.

....omissis.....

## > Screening

- Screening: Visit 1 (-12 weeks)

## > Randomization

- Randomization: Visit 2 (Day 1 +/- 5 days)

...omissis.....

| Visit | Day | Procedures/Assessments |
|---|---|---|
| Visit 1 | -12 Weeks | <ul> <li>Explanation to the patient of study aims, procedures and possible risks</li> <li>Informed consent signature</li> <li>Screening number</li> <li>Dispense patient card</li> <li>Demographic data and life style recording</li> <li>Medical/surgical history</li> <li>Previous/concomitant medications</li> <li>Full physical examination (weight, height, vital signs and physical abnormalities)</li> <li>Laboratory analyses: haematology, blood chemistry, urinalysis</li> <li>Evaluation of Inclusion/Exclusion criteria for eligibility</li> <li>Global Photograph</li> <li>Investigator &amp; blind assessor assessment</li> <li>AE monitoring</li> </ul> |
| Visit 2 | Day 1 | <ul> <li>Check concomitant medication</li> <li>Hair count macrophotography – baseline evaluation</li> <li>Global Photograph (if needed a reshoot)</li> <li>Inclusion/Exclusion criteria for eligibility</li> <li>Randomization</li> <li>Dispense study medication</li> <li>Dispense study diary</li> <li>AE monitoring</li> </ul> |

....omissis....

For all visits including global photo or hair count macrophotography, the patient may be asked to return to the site for reshoot if originally taken images are rejected by imaging vendor due to quality issues.

## 6.2 Investigator assessment

The local investigator will assess change in hair growth from baseline to Week 12 and from Baseline to Week 24, using a 7-point scale. The evaluation will be done by the Investigator or designee, by comparing the global vertex view photograph obtained at baseline screening visit with the patient's actual scalp at Week 12 and Week 24. This assessment will made separately based on changes to the vertex view. For the purpose of assessment of changes in hair growth by investigators and blind assessor screening visits (where global photos are taken) will act as Baseline. ...omissis.... 6.3 **Blind Assessor** ...omissis. This assessment will be performed by comparing the global photographs obtained at baseline screening visit with those subsequently obtained at Weeks 12 and 24. 7.2 Clinical laboratory assays Samples of blood (about 12.5 mL) and urine will be collected. The following laboratory analyses will be performed at Visits 1, 4 and 6 (ETV if applicable): 7.4 Total number of samples and blood withdrawn During the study, the following volume of blood will be collected: For routine laboratories analysis: Visit 1, 4 and 6, or at the ETV: 12-4.5 x 3 collections (excluding ETV: 4.5 ml) = about 37 13.5 mL In total, a maximum of about 121 55.5 mL of blood (not exceeding a normal blood donation) will be withdrawn from each patient during the entire study (about 28 30 weeks). 8.1.3 Route and method of administration

....omissis.....

After the application on clean, dry scalp, both topical solutions (P-3074 or its Vehicle) evaporate quickly leaving a water-permeable, transpirant transpiring, non-shining and almost invisible layer. ....omissis..... 8.1.4 Investigational product distribution All groups treatment kits will be provided by the investigator or by his/her deputy. They will be exclusively used for the present clinical study and will only be administered to the patients enrolled in the study. 8.2 Packaging and labelling The Sponsor will provide each site with individually treatment packs for each patient numbered treatment kits. ...omissis Each pack will be identified by a label bearing the frequency of administration, the treatment code and the number of bottles and tablets capsules contained; each label will be filled in with the site number, the randomization number and visit number by the Investigator 9.1.2 Secondary variables ...omissis.... Self-administered Male Hair Growth Questionnaire (MHGQ) score as assessed by the patient at Weeks 12 and 24 omissis.... 10.2.1 Analysis of Primary Efficacy Endpoint omissis The variance-covariance matrix of unstructured form will be used in order to model the correlation, within each patient, between the three two repeated measurements (over the post-baseline visits). omissis.... 10.2.2 Analysis of Secondary Efficacy Endpoints omissis • Self-administered Male Hair Growth Questionnaire (MHGQ) Score as assessed by the patient at Weeks 12 and 24

- Blind assessor assessment of patient hair growth/loss change from baseline: data will be fitted by a mixed linear model for repeated measures with treatment group, centre, visit and treatmentby-visit interaction as fixed effects, baseline value as covariate, and with an unstructured variance-covariance matrix to take into account correlations among repeated measures within patient. Results will be reported as maximum likelihood estimates of the treatment difference at Weeks 12 and 24 together with associated two-tailed 95% CI. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant.
- Change from baseline in Investigator Assessment at 12 and 24 weeks: data will be fitted by a mixed linear model for repeated measures with treatment group, centre, visit and treatment-byvisit interaction as fixed effects, baseline value as covariate, and with an unstructured variance-

covariance matrix to take into account correlations among repeated measures within patient. Results will be reported as maximum likelihood estimates of the treatment difference at Weeks 12 and 24 together with associated two-tailed 95% CI. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant.

| | Sample size and Power |
|---|---|
| | nissisature <sup>28,29</sup> shows that the mean change from baseline of hair count estimated in 1 inch <sup>2</sup> (= 6.25 |
| | · |
| | cm <sup>2</sup> ) and 1 cm <sup>2</sup> is correlated. For the above reason, the use of 1 inch <sup>2</sup> or 1 cm <sup>2</sup> , as vertex targ |
| | doesn't affect the sample size calculation. |
| on | nissis |
| 11.2 | Definitions |
| on | nissis |
| <b>→</b> | - events occurred after biopsies performed at Visit 2 (from day - 14 to day - 7) |
| on | nissis |
| 11.3 | AEs monitoring window |
| on | nissis |
| | E occurring after the follow up visit 7 (day 14±2 week 28) and coming to knowledge of the |
| inves | tigator (e.g. during a follow-up assessment or by spontaneous reporting by study patients) must be |
| recore | ded only if it is an ADR, according to the investigator's judgment. |
| 13 | References |
| on | nissis |
| <b>28.</b> | Gubelin Harcha W, Barboza Martínez J, Tsai TF, Katsuoka K, Kawashima M, Tsuboi R, |
| Barn | es A, Ferron-Brady G, Chetty D. A randomized, active- and placebo-controlled study of the |
| | ncy and safety of different doses of dutasteride versus placebo and finasteride in the ment of male subjects with androgenetic alopecia. J Am Acad Dermatol. 2014 |
| Mar; | 70(3):489-498. |
| <b>29.</b> | Blume-Peytavi U, Hillmann K, Dietz E, Canfield D, Garcia Bartels N. A randomized, |

single-blind trial of 5% minoxidil foam once daily versus 2% minoxidil solution twice daily in the treatment of androgenetic alopecia in women. J Am Acad Dermatol. 2011 Dec;65(6):1126-1134.